CLINICAL TRIAL: NCT03433053
Title: Developing Evidenced-Based Health Messages to Increase HIV Testing Among African-American Young Adult Women
Brief Title: Developing and Examining Evidenced-Based HIV Testing Messages
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HM20009273; 1F31MD011278-01A1 (NIH)
Record Dates: First submitted 2018-02-07; First posted 2018-02-14 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Participants will be exposed to a generic HIV testing message.
  Interventions: Behavioral: Control
- Experiment (Experimental): Participants will be exposed to a targeted HIV testing message, developed specifically for African American women.
  Interventions: Behavioral: HIV Testing Message Intervention

INTERVENTIONS:
Behavioral: HIV Testing Message Intervention — The Health Belief Model will be utilized as the primary theoretical framework in guiding the development of a tailored HIV testing message for young African American women in this intervention. Two conditions will be developed and compared as outlined below. Condition 1 participants will be exposed to an HIV testing message inclusive of culturally tailored information that addresses both culturally specific barriers and facilitators of HIV testing (as identified in Study 1). The message will be brief (will take less than 3 minutes to present/read).
  Arms: Experiment
Behavioral: Control — Condition 2 (generic message) participants will be exposed to a simple HIV educational message only, consisting of HIV statistics for women in the United States, information on how HIV is transmitted, where to get tested, and the benefits of HIV testing. The statistics on HIV and where to get tested will be taken directly from the CDC's website. The message will be brief (will take less than 3 minutes to present/read).
  Arms: Control

SUMMARY:
The goals of this study are to:

1. Develop a HIV test message tailored for African American women. A generic non-tailored message will be developed as well for comparison. A third group will be included that will not be exposed to any message at all.
2. Test the effectiveness of both messages on reported future intentions to get tested for HIV and HIV test behavior at 3 month follow up.

DETAILED DESCRIPTION:
African American women have the highest risk and prevalence of HIV infection among women of all racial/ethnic groups in the United States. Many of the current HIV infections among young adult African American women remain undiagnosed. The established benefits of routine HIV testing, the limitations of safer sex programs, and the gap of research related to increasing HIV testing as prevention necessitates the need for future research that specifically targets mechanisms to increase HIV testing. Higher rates of HIV testing can decrease rates of HIV transmission, as individuals who are knowledgeable of their status are less likely to transmit the virus. The current literature is sparse on factors related to HIV testing among young adults and has largely only examined demographic and sexual behavior correlates of HIV testing. Additionally, no studies have developed evidence-based health messages to promote HIV testing specifically among African American young women, despite their high risk of HIV infection and the importance of HIV testing. Thus, the proposed study will intend to identify factors related to HIV testing beyond the demographic and sexual risk level through formative research. These identified factors will be included as important elements in the development of HIV testing messages to motivate increased HIV testing. An enhanced message (culturally tailored) and a knowledge only message will be developed and tested.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified Black or African American women

Exclusion Criteria:

* Women who have never had sex, are married, or are pregnant/attempting to become pregnant

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 141 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2019-06-24 (Actual); Study Completion 2019-06-24 (Actual)

PRIMARY OUTCOMES:
HIV Test Intentions | Three month follow up
  Difference in future HIV test intentions between the tailored message group and the control group as measured by a follow up questionnaire, with higher scores indicating greater intention to be tested for HIV

CONTACTS AND LOCATIONS:
Overall Officials: Faye Belgrave, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States